CLINICAL TRIAL: NCT03862170
Title: Antibiotic Prophylaxis for HDR Brachytherapy in the Treatment of Prostate Cancer: a Phase III Randomized Trial
Brief Title: Antibiotic Prophylaxis for HDR Brachytherapy in the Treatment of Prostate Cancer
Acronym: BRP30
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Covid-19 pandemic
Sponsor: CR-CSSS Champlain-Charles-Le Moyne (Other)
Responsible Party: Principal Investigator, Marjory Jolicoeur, Principal Investigator, MD, PhD, CR-CSSS Champlain-Charles-Le Moyne
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AA-HCLM-14-033
Record Dates: First submitted 2018-06-28; First posted 2019-03-05 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Prostate Cancer
Keywords: HDR Brachytherapy; prophylactic antibiotics; ciprofloxacin; ancef; RCT
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Ciprofloxacin; Cefazolin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ciprofloxacin (Active Comparator): Patients in this arm will receive Ciprofloxacin 400mg IV 120mn (prophylactic antibiotic) before their HDR brachytherapy
  Interventions: Drug: Ciprofloxacin
- Cefazolin (Experimental): Patients in this arm will receive Cefazolin 2000mg IV 60mn (prophylactic antibiotic) before their HDR brachytherapy
  Interventions: Drug: Cefazolin
- No prophylactic antibiotics (No Intervention): Patients in this arm will not receive any prophylactic antibiotics before their HDR brachytherapy

INTERVENTIONS:
Drug: Ciprofloxacin — Ciprofloxacin 400 mg IV 120mn before HDR brachytherapy
  Other Names: Ciloxan; Cipro; Neofloxin
  Arms: Ciprofloxacin
Drug: Cefazolin
  Other Names: Ancef; cefazoline; cephazolin; Cefacidal
  Arms: Cefazolin

SUMMARY:
Phase III study that aims to evaluate the necessity of prophylactic antibiotics use after HDR brachytherapy in the treatment of prostate adenocarcinomas.

DETAILED DESCRIPTION:
INTRODUCTION:

High dose rate (HDR) brachytherapy boost with external beam is the current recommended treatment for intermediate and high risk prostate cancers (1, 2). HDR brachytherapy uses transperineal implant (at least 15 prostate catheters) to deliver the calculated dose though a robot that contains the radioactive source. Once treatment is completed, the implant is retrieved and a dressing with an antibiotic ointment is placed on the perineum for a few hours.

The procedure is performed under spinal anesthesia, transperineally following a sterile wash. The implantation is guided from the transrectal ultrasound (TRUS). The procedure contains a series of back and forth probe movements that raises the contamination risk of the implantation zone which is considered non-negligible. Brachytherapy patients undergo urinanalysis before the implantation and redo the test at the least urinary symptom.

The suspicion of a contamination risk of the urinary tract during the procedure has therefore led to antibiotic prophylaxis habit. This habit has been based on experts' opinion mainly motivated by the antibiotic prophylaxis use for TRUS guided biopsies of the prostate.

Literature on antibiotic prophylaxis use for prostate brachytherapy is limited, both on the use of intraoperative or post-procedure antibiotic prophylaxis and on the risk of infectious complications following the brachytherapy procedure.

The use of antibiotic prophylaxis for prostate brachytherapy is derived from urology studies based on prostate biopsies (3, 4). Nevertheless, biopsy procedure is completely different from the implantation used on brachytherapy. Moreover, biopsies are done transrectally with bacterial dissemination risk on blood circulation, while brachytherapy is done transperineally.

Current recommendations from American Brachytherapy Society (ABS) do not state on the use of antibiotic prophylaxis for brachytherapy prostate patients (5). Antibiotic prophylaxis is however cited as possibly useful. The European Society for Radiation and Oncology (GEC-ESTRO) does not comment on the need for antibiotic prophylaxis, but mentions cystitis as a possible complication for prostate brachytherapy (1, 2). It is important to consider that these recommendations are based on expert opinion (level of evidence V). Unfortunately, there is no randomized trial (level of evidence I) to guide the use of antibiotic prophylaxis for prostate brachytherapy.

The most current used molecule for the antibiotic prophylaxis of the urinary tract is Ciprofloxacin. Yet, Ciprofloxacin is linked to the upsurge of C. difficile and the use of this molecule is linked to the appearance of many bacterial strains resistant to antibiotics (6). Other antibiotics, like Cefazolin do not have the same association with C. difficile and other multidrug-resistant bacteria. Cefazolin is equally used as antibiotic prophylaxis for pelvic surgery. Investigators can suppose that Ciprofloxacin can be replaced by Cefazolin as an antibiotic prophylaxis for prostate brachytherapy, causing less harm.

Moreover, one study compared both antibiotics (Ciprofloxacin and Cefazolin) in the prophylactic use in 100 patients (7). Authors demonstrated equivalence between both drugs for the prevention of urinary contamination. Although the study was not designed to demonstrate equivalence and the observed effect may be due to low number of randomized patients.

Furthermore, this study has not demonstrated beyond any doubt the need of antibiotic prophylaxis for prostate brachytherapy. Investigators continue to be uncertain about the need of antibiotic prophylaxis, as the rate of urinary infections without antibiotic prophylaxis after prostate brachytherapy continues to be unknown.

Nevertheless, radiation side effects on the urinary function are well known and are systematically reviewed by validate questionnaires, such as International Prostate Symptom Score (IPSS) and are graded accordingly to the Common Terminology Criteria for Adverse Events (CTCAE) score.

In summary, there is no evidence in the literature of the need for antibiotic prophylaxis in prostate brachytherapy. Likewise, there is no evidence to support that if used, it should be Ciprofloxacin. Furthermore, in times of multidrug-resistant bacteria, it is important to decrease the use of these molecules. This is why the investigators propose a phase III randomized clinical trial to evaluate the risk of urinary tract infection in the presence or absence of antibiotic prophylaxis for prostate brachytherapy.

METHODS:

Hypothesis:

The investigators hypothesize that the risk of infectious complication of the urinary tract following prostate brachytherapy is the same with or without antibiotic prophylaxis.

Objectives:

Primary:

- Evaluate the rate of urinary tract infections following prostate brachytherapy.

Secondary:

* Evaluate the rate and grade of the urinary tract complications in the presence and absence of antibiotics.
* Evaluate the effect on the IPSS score in the presence and absence of antibiotics.
* Evaluate the rate of serious infectious complications related to brachytherapy.
* Evaluate the risk of colitis due to C. difficile in the 12 weeks following the brachytherapy

Patient selection:

Inclusion and exclusion criteria are described elsewhere.

Pre-implant evaluation (morning of the intervention):

* Urinary test and culture
* Bladder scan

Treatment:

The patients are treated by HDR brachytherapy boost with external beam according to the current standards. Current standard also premise that patients are followed up weekly by their doctor. During patient visits, urinary symptoms questionnaire is fulfilled and urinary tests are performed as needed.

In the study establishment, patient is seen the next day of the procedure to retrieve the urinary catheter left after the procedure. During this visit a bladder scan post-miction is performed to check the bladder residual volume.

Antibiotic prophylaxis:

Randomization in 3 arms: Ciprofloxacin 400 mg IV 120 mn pre-operative, Cefazolin 2g IV 60 mn pre-operative or no antibiotic prophylaxis.

Data gathering:

Patient is to be seen day of the procedure (day 0), the next day (day 1), 3 days after the procedure (day 3), one week after (day 7), 1 month (day 30) and 3 months after procedure (day 90). Patients will fulfill IPSS questionnaire, make urine tests and a bladder scan in every visit.

Patients will be seen weekly during the external beam treatment by their doctor. Patient's symptoms will be graded according to the RTOG score. In cases with suspicion of urinary tract infection or prostatitis during the treatments, the standard procedure with urinary tests will take place.

Statistical Analysis:

The basic assumption is the probability of no difference in bacteriuria and change in the IPSS score between the 3 arms.

Sample size:

A difference of 15% between the groups equates to an effect size of 0.24 which is the magnitude of Chi-square that needs to be detected, gives us a power of 83%. Calculation was done using the PASS software.

A total of 234 eligible patients (78 per arm) are required for a power of 92% and a risk of the first species of 0.05. Adjust for 10% of ineligibility, the number needed is 255 patients (85 per arm).

Data analysis :

Data reading and statistical analysis will be done by the Statistical Analysis Software (SAS) package.

Socio-demographic characteristics, IPSS scores and patient's clinical data will be described by descriptive statistics (means, standard deviation, proportions, etc.). Anova or Chi-square tests will be used to compare arms. Multivariate logistic regression models will allow us to determine the potential associations between our categorical dependent variables while controlling for both sociodemographic factors and especially for potentially confounding clinical variables.

ELIGIBILITY:
Inclusion Criteria:

* All patients eligible to brachytherapy for the treatment of prostate cancer
* No history of serious urinary tract infection post prostate biopsy

Exclusion Criteria:

* Urosepsis post biopsy
* Contraindication to brachytherapy

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2015-02-10 (Actual); Primary Completion 2020-02 (Actual); Study Completion 2023-02 (Actual)

PRIMARY OUTCOMES:
Symptomatic urinary infections post HDR brachytherapy | from treatment up to 6 months, divided into acute (up to 3 months post treatment) and late (between 3 and 6 months post treatment)
  The rate of symptomatic urinary infections post HDR brachytherapy.

SECONDARY OUTCOMES:
Urinary toxicities | 5 years
  Urinary toxicities rate in each arm measured by the Common Terminology Criteria for Adverse Events (CTCAE) score. The following Medical Dictionary for Regulatory Activities (MedDRA) System Organ Classes (SOC) will be included: Renal and urinary disorders, and Infections and infestations. The CTCAE score ranges from grade 0 to 5, where higher grade represents higher toxicity. Each presented toxicity will be assessed and scored. Each toxicity will be evaluated by its percentage of incidence in the sample. Each patient will also be evaluated by his worse toxicity (higher grade). The percentage of toxicities incidence and their severity will be compared between groups.
IPSS score effects | 5 years
  Evaluate International Prostate Symptom Score (IPSS) effects of prophylactic antibiotics. The IPSS Score ranges from 0 to 35. A score of 0 to 7 indicates mild symptoms, 8 to 19 indicates moderate symptoms and 20 to 35 indicates severe symptoms. Mean scores will be compared between groups.
Serious infectious complications | 5 years
  Evaluate the rate of serious infectious complications post HDR brachytherapy
The risk of colitis due to C. difficile infection | 12 weeks
  To evaluate the risk of colitis due to C. difficile infection all patients with diarrhea or increased bowel movement (colitis symptoms) will be tested for C. difficile infection. The association between colitis and the presence of C. difficile infection will be evaluated by Chi-square in each group.

CONTACTS AND LOCATIONS:
Overall Officials: Marjory Jolicoeur, MD,MSc, Principal Investigator — CSSS Champlain-Charles-Le Moyne
Locations (1):
- Hôpital Charles LeMoyne, Greenfield Park, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kovacs G, Potter R, Loch T, Hammer J, Kolkman-Deurloo IK, de la Rosette JJ, Bertermann H. GEC/ESTRO-EAU recommendations on temporary brachytherapy using stepping sources for localised prostate cancer. Radiother Oncol. 2005 Feb;74(2):137-48. doi: 10.1016/j.radonc.2004.09.004. PMID 15734201
- [Background] Hoskin PJ, Colombo A, Henry A, Niehoff P, Paulsen Hellebust T, Siebert FA, Kovacs G. GEC/ESTRO recommendations on high dose rate afterloading brachytherapy for localised prostate cancer: an update. Radiother Oncol. 2013 Jun;107(3):325-32. doi: 10.1016/j.radonc.2013.05.002. Epub 2013 Jun 14. PMID 23773409
- [Background] Puig J, Darnell A, Bermudez P, Malet A, Serrate G, Bare M, Prats J. Transrectal ultrasound-guided prostate biopsy: is antibiotic prophylaxis necessary? Eur Radiol. 2006 Apr;16(4):939-43. doi: 10.1007/s00330-005-0076-2. Epub 2006 Jan 4. PMID 16391904
- [Background] Griffith BC, Morey AF, Ali-Khan MM, Canby-Hagino E, Foley JP, Rozanski TA. Single dose levofloxacin prophylaxis for prostate biopsy in patients at low risk. J Urol. 2002 Sep;168(3):1021-3. doi: 10.1016/S0022-5347(05)64565-X. PMID 12187213
- [Background] Yamada Y, Rogers L, Demanes DJ, Morton G, Prestidge BR, Pouliot J, Cohen GN, Zaider M, Ghilezan M, Hsu IC; American Brachytherapy Society. American Brachytherapy Society consensus guidelines for high-dose-rate prostate brachytherapy. Brachytherapy. 2012 Jan-Feb;11(1):20-32. doi: 10.1016/j.brachy.2011.09.008. PMID 22265435
- [Background] Deshpande A, Pant C, Jain A, Fraser TG, Rolston DD. Do fluoroquinolones predispose patients to Clostridium difficile associated disease? A review of the evidence. Curr Med Res Opin. 2008 Feb;24(2):329-33. doi: 10.1185/030079908x253735. PMID 18067688
- [Background] Christiano AP, Hollowell CM, Kim H, Kim J, Patel R, Bales GT, Gerber GS. Double-blind randomized comparison of single-dose ciprofloxacin versus intravenous cefazolin in patients undergoing outpatient endourologic surgery. Urology. 2000 Feb;55(2):182-5. doi: 10.1016/s0090-4295(99)00412-4. PMID 10688075